CLINICAL TRIAL: NCT05918315
Title: Dorsolateral Versus Dorsal Approach Urethroplasty for Managing Long Anterior Urethral Stricture.
Brief Title: Comparison Between Two Techniques Used in Treatment of Long Anterior Urethral Stricture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hosny Fathallah Omar, MD, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-06-01MD
Record Dates: First submitted 2023-06-14; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Urethral Stricture, Male
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dorsolateral approach urethroplasty (Active Comparator): Use of dorsolateral(Kulkarni technique) urethroplasty.
  Interventions: Procedure: Buccal mucosa substitution urethroplasty
- Dorsal approach urethroplasty (Active Comparator): Use of dorsal (Barbagli technique) urethroplasty
  Interventions: Procedure: Buccal mucosa substitution urethroplasty

INTERVENTIONS:
Procedure: Buccal mucosa substitution urethroplasty — Use of buccal mucosa as a substitution for urethroplasty

SUMMARY:
To evaluate dorsolateral and dorsal approach urethroplasty in treatment of anterior urethral stricture by using buccal mucosal graft as regard voiding and sexual outcomes.

DETAILED DESCRIPTION:
At the Department of Urology, Sohag university Hospital, both techniques of dorsolateral and dorsal approach urethroplasty in treatment of anterior urethral stricture by using buccal are used in repair of long stricture anterior urethra.Therefore, our data can be used as a source for the comparative analysis of these two Buccal mucosa graft urethroplasty techniques.This study aimed to compare these procedures to determine their advantages and disadvantages, as regard voiding ,sexual function and quality of life after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* long anterior urethral stricture

Exclusion Criteria:

* children.
* Recurrent stricture

Ages: 16 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Voiding function | 2 months after catheter removal
  Postoperative Q max

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Reyad, MD, Study Director — Sohag University
Locations (1):
- Sohag university, Sohag, Faculty of Medicine, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Share collected IPD
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months after publication